CLINICAL TRIAL: NCT05779449
Title: Targeting the Gut Dysbiosis to Treat Inflammation-driven Synaptopathy in Multiple Sclerosis
Brief Title: Targeting the Gut Dysbiosis to Treat Inflammation-driven Synaptopathy in MS
Acronym: Pre-Pro-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Collaborators: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Diego Centonze, Head of Neurology Unit, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pre-Pro-MS
Record Dates: First submitted 2023-03-06; First posted 2023-03-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Patient Participation
Keywords: gut microbiota; dysbiosis; multiple sclerosis; glutamate-mediated excitotoxicity; synaptopathy
MeSH Terms: conditions — Patient Participation; Dysbiosis; Multiple Sclerosis | interventions — Prebiotics; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Pro group (Experimental): Patients with RRMS under dimethyl fumarate or Ocrelizumab treatment according to the good clinical practice, who will recieve the following dietary supplementation with pre- and probiotics:
  1st-15th days: One capsule containg 6 billions of Saccharomyces boulardii and 8,5 billions of probiotics including Bifidobacterium lactis Bi-07®, Bifidobacterium lactis Bl-04, Lacticaseibacillus paracasei Lpc-37, Lactobacillus acidophilus NCFM® (Probactiol Duo cps, Metagenics) One packet with 4 g of prebiotics including inulin enriched with oligofructose (Probactiol Stips bustine Metagenics).
  16th-365th days:
  Two capsules, each containg 7,5 billions of Lactobacillus acidophilus NCFM®, 7,5 billions of Bifidobacterium lactis Bi-07®, 2,5 ug Vitamine D3, 320 ug Vitamine A, 100 mg Threonine, 250 mg 2'-Fucosyllactose (Probactiol HMO Combi cps, Metagenics).
  Interventions: Dietary Supplement: Prebiotics and Probiotics supplementation; Procedure: peripheral blood withdrawal; Procedure: Transcranial Magnetic Stimulation (TMS)
- Placebo group (Placebo Comparator): Patients with RRMS under dimethyl fumarate or Ocrelizumab treatment according to the good clinical practice, who will receive only starch, the probiotic bacteria carrier:
  1st-15th days: One capsule and one packet only with starch.
  16th-365th days: Two capsules containg starch.
  Interventions: Dietary Supplement: Placebo supplementation; Procedure: peripheral blood withdrawal; Procedure: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Dietary Supplement: Prebiotics and Probiotics supplementation — From the 1st day to the 15th day (included) patients with MS in the Pre-Pro group will receive daily:
  1 capsule of Probactiol Duo, Metagenics (6 billions of Saccharomyces boulardii and 8,5 billions of probiotics including Bifidobacterium lactis Bi-07®, Bifidobacterium lactis Bl-04, Lacticaseibacillus paracasei Lpc-37, Lactobacillus acidophilus NCFM®)
  1. packet of Probactiol Stips, Metagenics (4 g inulin enriched with oligofructose)
     From the16th day to the 365th day (included) patients with MS in the Pre-Pro group will receive daily:
  2. capsules of Probactiol HMO Combi, Metagenics (7,5 billions of Lactobacillus acidophilus NCFM®, 7,5 billions of Bifidobacterium lactis Bi-07®, 2,5 ug Vitamine D3, 320 ug Vitamine A, 100 mg Threonine, 250 mg 2'-Fucosyllactose).
  Arms: Pre-Pro group
Dietary Supplement: Placebo supplementation — 1-year supplementation with two placebo capsules/day containing starch, the probiotic bacteria carrier.
  Arms: Placebo group
Procedure: peripheral blood withdrawal — 40 ml of blood for the isolation of Peripheral Blood Cells (PBMCs) and T cells.
Procedure: Transcranial Magnetic Stimulation (TMS) — Intermittent theta burst stimulation (iTBS) protocol

SUMMARY:
Inflammatory synaptopathy is a prominent pathogenic process in multiple sclerosis (MS) induced by imbalanced immune system homeostasis. Its persistence causes excitotoxic neuronal damage, leading to motor and cognitive deficits. Although many advances have been made in MS treatment, the development of effective strategies for managing disease progression driven by excitotoxic synaptic dysfunctions is of great significance. Gut dysbiosis is commonly associated with both MS and obesity and high-fat diet (HFD) can exacerbate disease by acting on gut microbiota.

Since gut microbiota can shape the immune response and brain functions, we propose to target gut dysbiosis by dietary supplementation of prebiotics and probiotics (Pre-Pro) to treat synaptopathy in both human and experimental model of MS, even when exacerbated by HFD. Overall, this project aims at unveiling the anti-inflammatory and neuroprotective pathways activated by Pre-Pro supplementation to modulate the immune-synaptic axis.

DETAILED DESCRIPTION:
MS is a chronic autoimmune neurodegenerative disease characterized by different forms. The most common is the relapsing-remitting (RR)MS showing a significant dysregulation of immune homeostasis.

Disease progression occurring during MS, is not only driven by infiltrating T cells destroying myelin during relapses, indeed proinflammatory molecules can also trigger a glutamate-induced excitotoxic synaptopathy promoting neurodegenerative processes and negatively influencing disease course.

Inflammation, synaptopathy and neurodegeneration are intermingled with reparative processes in different proportions, making the MS course unpredictable and the treatment approach challenging. Lifestyle habits can contribute to the heterogeneity of MS pathophysiology. In this context, the gut microbiota is emerging as a key sensor of lifestyle indeed it is continuously modulated by many factors, particularly dietary habits, and by controlling the immune system homeostasis can influence the onset and progression of MS.

HFD exacerbates MS by promoting neuroinflammation and affects gut microbiota inducing dysbiosis.

Gut dysbiosis in MS is associated with increased microglia activation and imbalance between pathogenic Th1/Th17 and tolerogenic regulatory T (Treg cells), however its effects on immune-mediated synaptopathy and their underlying mechanisms in MS have not yet been investigated.

Considering that excitotoxic synaptic dysfunctions are reversible and can be only partially controlled by the currently available disease-modifying treatments (DMTs), they represent an attractive therapeutic target in MS. Microbiota manipulation by dietary prebiotics and probiotics (Pre-Pro) supplementation may be an attractive candidate for enhancing the efficacy and the anti-synaptotoxic action of DMTs and could result in a safer and more effective therapeutic strategy to improve the management of overall health and well-being of MS patients.

This clinical study will be performed to verify whether the gut-microbiota manipulation can counteract synaptic alterations, neuroinflammation and degeneration by switching the immune system towards a more tolerogenic phenotype thus improving MS cognitive and clinical outcomes.

To verify our hypothesis, we will perform clinical and experimental studies to dissect at cellular and molecular level the effect and the mechanism of action of Pre-Pro supplementation during MS.

The following objectives will be addressed by evaluating the effects of a dietary supplementation of prebiotics and probiotics (Pre-Pro) in RRMS patients on

1. clinical disability and disease course;
2. immune cell homeostasis;
3. inflammation-driven synaptopathy and its molecular determinants.

This project aims at investigating for the first time the impact of gut-microbiota modulation on MS course associated with excitotoxic synaptopathy. The multidisciplinary approach will provide the unique opportunity to dissect immunoregulatory and synaptic effects of the prolonged Pre-Pro intake at both cellular and molecular levels. Moreover, the possible identification of novel molecular actors controlling the immune-brain axis shaped by the microbiota will open new opportunities for expanding the current treatment options for MS.

Overall, the results of this project will provide robust scientific groundwork for an integrative medicine based on Pre-Pro supplementation in addition to first line drug treatments for MS to counteract synaptopathy-driven disease progression.

ELIGIBILITY:
Inclusion Criteria:

* RRMS diagnosis, as Polman et al 2011. Ann Neurol. PMID: 21387374
* Age <= 18 and => 65 years
* EDSS score <= 7
* Disease duration < 10 years
* On DMF or Ocrelizumab treatment from at least 3 months
* No corticosteroid administration in the previous month
* Ability to provide written informed consent.

Exclusion Criteria:

* Adverse effects to gadolinium
* Blood count basal alteration
* Pregnant or lactating women
* Vegetarians or vegans
* Taking antibiotics, any product or supplement containing probiotics, Omega 3 or other antioxidant supplements within 30 days prior to inclusion
* History of food allergies or food intolerance
* Clinically significant medical condition other than MS, (latent infections, other autoimmune disease)
* Diagnosis of past eating disorders (anorexia, bulimia, or binge eating) or relevant psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-11-02 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota diversity or composition | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Relative taxa abundance in fecal samples assessed by rDNA-seq (Operational Taxonomy Unit, OTU).
Changes in microbiota metabolites - indican | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Quantification of the ration between indican and creatinine (μg/mg) in urine samples
Changes in microbiota metabolites - skatole | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Quantification of the ration between skatole and creatinine (μg/mg) in urine samples
Changes in serum glutamate | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Absolute quantification of glutamate in the serum (uM)
Changes in serum synaptotoxic miRNAs | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Relative quantification by Real-time PCR
Changes in plasma inflammatory molecules | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Absolute quantification of inflammatory molecules in the serum (pg/ml)
Changes in immunophenotype | T0 vs T12 (months), Pre-Pro versus Placebo groups
  The percentage of Treg in the activated CD4+CD25- T cells isolated from PMBCs will be evaluated by Fluorescence-activated Cell Sorting (FACS).
Changes in T cell metabolic asset | T0 vs T12 (months), Pre-Pro versus Placebo groups
  The metabolic profile of CD4+ T cells will be assessed by real-time measurement of extracellular acidification rate (ECAR) and oxygen consumption rate (OCR), using an XFe-96 Extracellular Flux Analyzer.

SECONDARY OUTCOMES:
Changes in neurophysiological response | T0 vs T12 (months), Pre-Pro versus Placebo groups
  A protocol of Intermittent theta burst stimulation (iTBS) will be used to evaluate change in Motor-Evoked Potentials (MEP) before (baseline) and after 15 and 30 minutes from stimuli (10 bursts, each burst composed of three stimuli at 50 Hz).
  Twenty MEPs will be collected at each time points.MEP's amplitudes will be averaged at each time point and normalized to the mean baseline amplitude.
Changes in clinical disability | T0 vs T12 (months), Pre-Pro versus Placebo groups
  The Expanded Disability Status Scale (EDSS)/Kurtzke is widely used in MS clinical pactice and trials to quantify disability and monitor the changes in the level of disability over time. The EDSS scale ranges from 0 to 10.
Changes in lower extremity function | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Quantitative measure of lower extremity function will be performed by the Timed 25-Foot Walk (T25FW). The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The average score of two 25-Foot Timed Walk trials will be measured.
Changes in upper extremity function | T0 vs T12 (months), Pre-Pro versus Placebo groups
  The upper extremity (arm and hand) function will be assessed by 9-Hole Peg Test (9HPT). Both the dominant and non-dominant hands are tested twice. Two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand will be executed.
Changes in quality of life | T0 vs T12 (months), Pre-Pro versus Placebo groups
  The Multiple Sclerosis Quality of Life-54 (MSQOL-54) is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument.
  The test includes 36 items as the generic component and 18 items added to tap MS-specific issues such as fatigue, cognitive function, etc. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The summary scores are the physical health composite summary and the mental health composite summary. The single item measures are satisfaction with sexual function and change in health.
  Administration time of this structured, self-report questionnaire is approximately 11-18 minutes.
Assessment of mild to moderate dysfunctions | T0 vs T12 (months), Pre-Pro versus Placebo groups
  The Paced Auditory Serial Addition Test (PASAT) will be used to measure the cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The score for the PASAT is the total number correct out of 60 possible answers. This score can be used individually or used as part of the MSFC composite score. Administration time is approximately 10-15 minutes including practice sessions.
Changes in global cognitive disability | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Mini Mental State Examination (MMSE) will be used to assess cognitive function including orientation, attention, memory, language and visual-spatial skills.
Assessment of attention and information processing speed | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Attention and information processing speed will be evaluated by the Symbol Digit Modality Test (SDMT).
  The examinee has 90 seconds to pair specific numbers with given geometric figures by using a reference key. The SDMT score is the sum of the correct substitutions within the 90 second interval.
Changes in phonemic verbal fluency | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Word List Generation (WLG) will be used as a phonemic verbal fluency task to evaluate the spontaneous production of words and mental flexibility, when given a letter from the alphabet and within a limited amount of time (one minute).
Changes in verbal memory performance | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Rey Auditory Verbal Learning Test (RAVLT) will be used to evaluate verbal memory.
Changes in measure visuospatial memory | T0 vs T12 (months), Pre-Pro versus Placebo groups
  The Brief Visuospatial Memory Test-Revised (BVMT-R) will be used to measure visuospatial memory.
Changes in depressive symptoms | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Beck Depression Inventory-Second Edition (BDI-II) will be used to assess the presence of depressive symptoms. This scale includes 21 items and investigates both somatic and cognitive-affective symptoms, the score range is from 0 to 63. A cutoff of 13 will be used to detect depression.
Changes in anxious symptoms | T0 vs T12 (months), Pre-Pro versus Placebo groups
  State-Trait Anxiety Inventory form Y (STAI-Y) will be used to asses levels of anxiety. It consists of a 40-item self-administered questionnaire exploring both the levels of situational anxiety (state) and the tendency to anxious situations (trait). A cutoff for high anxiety will be derived according to normative data.
Changes in disease progression index (PI) | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Progression index (PI) is the ratio between EDSS (Expanded Disability Status Scale) and disease duration in months.
Changes in the Annualized Relapse Rate (ARR) | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Change in Annualized Relapse Rate (ARR) measured by the total number of relapses divided by the total person-time at risk of relapse.
Changes in radiological activity | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Radiological activity will be evaluated by conventional MRI scans (1.5 Tesla) after intravenous gadolinium (Gd) infusion (0.2 ml/kg). An active scan is defined as showing any new, enlarging or recurrent lesion(s) on T1-weighted spin-echo images (T1-WI) and T2-weighted spin-echo images (T2-WI).
  A new Gd+ lesion is defined as a typical area of hyperintense signal on postcontrast T1-WI.
  A new or newly enlarging lesion on T2-WI is defined as a rounded or oval lesion arising from an area previously considered as normal appearing brain tissue and/or showing an identifiable increase in size from a previously stable-appearing lesion.
Changes in brain atrophy | T0 vs T12 (months), Pre-Pro versus Placebo groups
  Difference of cortical thickness, the volume of subcortical grey matter structures and lesion volume will be evaluated by MRI scan

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS INM-Neuromed, Pozzilli, Isernia, Italy

REFERENCES:
- [Background] Mandolesi G, Gentile A, Musella A, Fresegna D, De Vito F, Bullitta S, Sepman H, Marfia GA, Centonze D. Synaptopathy connects inflammation and neurodegeneration in multiple sclerosis. Nat Rev Neurol. 2015 Dec;11(12):711-24. doi: 10.1038/nrneurol.2015.222. Epub 2015 Nov 20. PMID 26585978
- [Background] De Vito F, Musella A, Fresegna D, Rizzo FR, Gentile A, Stampanoni Bassi M, Gilio L, Buttari F, Procaccini C, Colamatteo A, Bullitta S, Guadalupi L, Caioli S, Vanni V, Balletta S, Sanna K, Bruno A, Dolcetti E, Furlan R, Finardi A, Licursi V, Drulovic J, Pekmezovic T, Fusco C, Bruzzaniti S, Hornstein E, Uccelli A, Salvetti M, Matarese G, Centonze D, Mandolesi G. MiR-142-3p regulates synaptopathy-driven disease progression in multiple sclerosis. Neuropathol Appl Neurobiol. 2022 Feb;48(2):e12765. doi: 10.1111/nan.12765. Epub 2021 Oct 6. PMID 34490928
- [Background] Stampanoni Bassi M, Iezzi E, Buttari F, Gilio L, Simonelli I, Carbone F, Micillo T, De Rosa V, Sica F, Furlan R, Finardi A, Fantozzi R, Storto M, Bellantonio P, Pirollo P, Di Lemme S, Musella A, Mandolesi G, Centonze D, Matarese G. Obesity worsens central inflammation and disability in multiple sclerosis. Mult Scler. 2020 Sep;26(10):1237-1246. doi: 10.1177/1352458519853473. Epub 2019 Jun 4. PMID 31161863
- [Background] Buckman LB, Hasty AH, Flaherty DK, Buckman CT, Thompson MM, Matlock BK, Weller K, Ellacott KL. Obesity induced by a high-fat diet is associated with increased immune cell entry into the central nervous system. Brain Behav Immun. 2014 Jan;35:33-42. doi: 10.1016/j.bbi.2013.06.007. Epub 2013 Jul 4. PMID 23831150
- [Background] Haase S, Wilck N, Haghikia A, Gold R, Mueller DN, Linker RA. The role of the gut microbiota and microbial metabolites in neuroinflammation. Eur J Immunol. 2020 Dec;50(12):1863-1870. doi: 10.1002/eji.201847807. Epub 2020 Dec 7. PMID 33188704
- [Background] Mirashrafi S, Hejazi Taghanaki SZ, Sarlak F, Moravejolahkami AR, Hojjati Kermani MA, Haratian M. Effect of probiotics supplementation on disease progression, depression, general health, and anthropometric measurements in relapsing-remitting multiple sclerosis patients: A systematic review and meta-analysis of clinical trials. Int J Clin Pract. 2021 Nov;75(11):e14724. doi: 10.1111/ijcp.14724. Epub 2021 Aug 19. PMID 34379879
- [Background] Siracusa F, Schaltenberg N, Villablanca EJ, Huber S, Gagliani N. Dietary Habits and Intestinal Immunity: From Food Intake to CD4+ T H Cells. Front Immunol. 2019 Jan 15;9:3177. doi: 10.3389/fimmu.2018.03177. eCollection 2018. PMID 30697217
- [Background] Valizadeh S, Majdi Seghinsara A, Maleki Chollou K, Bahadori A, Abbaszadeh S, Taghdir M, Behniafar H, Riahi SM. The efficacy of probiotics in experimental autoimmune encephalomyelitis (an animal model for MS): a systematic review and meta-analysis. Lett Appl Microbiol. 2021 Oct;73(4):408-417. doi: 10.1111/lam.13543. Epub 2021 Aug 11. PMID 34310737
- [Background] Sichetti M, De Marco S, Pagiotti R, Traina G, Pietrella D. Anti-inflammatory effect of multistrain probiotic formulation (L. rhamnosus, B. lactis, and B. longum). Nutrition. 2018 Sep;53:95-102. doi: 10.1016/j.nut.2018.02.005. Epub 2018 Feb 14. PMID 29674267